CLINICAL TRIAL: NCT06768723
Title: Effects of Post-activation Performance Enhancement Protocols Using Upper-body, Lower-body, or Combined Upper- and Lower-body Exercises on Judo-specific Performance: a Randomized Crossover Trial
Brief Title: Effects of Post-activation Performance Enhancement Protocols on Judo-specific Performance: a Randomized Crossover Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade do Porto (Other)
Collaborators: Rashtriya Raksha University (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: IRB/SPES/NOC/2023-24/03
Record Dates: First submitted 2025-01-06; First posted 2025-01-10 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: No Condition, Basic Science
Keywords: PAPE; Judo; Warm-Up
MeSH Terms: interventions — Warm-Up Exercise

STUDY DESIGN:
Intervention Model Description: A randomized crossover research design was used to analyze the effects of three PAPE-aimed conditioning exercises on the SJFT performance. The participants attended a total of five sessions during the study. The first session was used to familiarize the participants with the PAPE-aimed conditioning exercises. The participants had previous experience with the SJFT; however, the protocol was re-explained and performed by the participants during the familiarization session. The use of the RPE scale was also explained during this session, and demographic data were collected. Participants performed the three experimental protocols (i.e., combined, upper-body, lower-body) and the control condition (i.e., judo-specific warm-up) in four separate sessions (≥48 hours of recovery between sessions) in random order. All the testing sessions were conducted between 1400 and 1600 hours with an environmental temperature of approximately 28° C.
Who Masked: Outcomes Assessor
Masking Description: Assessors unknowing of the allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Upper body PAPE protocol (Experimental): Half of the judo-specific protocol + 3 sets of 10-second hold isometric push-ups.
  Interventions: Other: Warm-up (specifically, Post-Activation Performance Enhancement)
- Lower body PAPE protocol (Experimental): Half of the judo-specific protocol + 3 sets of 6 repetitions of standing broad jump.
  Interventions: Other: Warm-up (specifically, Post-Activation Performance Enhancement)
- Combined (Upper body+Lower body) PAPE protocol (Experimental): Half of the judo-specific protocol + 3 sets of 3 repetitions of standing broad jump + 3 sets of 5-second hold isometric push-ups.
  Interventions: Other: Warm-up (specifically, Post-Activation Performance Enhancement)
- Control (judo-specific) protocol (Active Comparator): Judo-specific exercises that included 10 repetitions of ukemi drills (i.e., front, back, side, and rolling), 2 sets of 10 repetitions of "rapid" uchikomi drills (i.e., throwing drills), 2 sets of 1 minute of kumikata fight (i.e., grip fight), and 2 sets of 10 repetitions of nagekomi (i.e., practice throws).
  Interventions: Other: Warm-up (specifically, Post-Activation Performance Enhancement)

INTERVENTIONS:
Other: Warm-up (specifically, Post-Activation Performance Enhancement) — Assess which intervention delivered the best acute performance enhancements.

SUMMARY:
The study aimed to investigate the post-activation performance enhancement (PAPE) of the special judo fitness test (SJFT) of youth judo athletes using upper-body (isometric push-ups), lower-body (standing broad jumps), or their combination as conditioning exercise (CE).

DETAILED DESCRIPTION:
Fourteen females (aged 16.5 ± 0.8 yrs) and nine males (aged 17.0 ± 0.9 yrs) performed the three CEs or a control condition (i.e., judo-specific warm-up) in a randomized crossover method. The SJFT was conducted one minute after the CE or control condition.

ELIGIBILITY:
Inclusion Criteria:

* Minimum of 4 years of judo training and competition experience.
* Actively practicing the sport and preparing for a competition during the time of data collection
* Proficient at performing the ippon seoi-nage throwing (judo) technique

Exclusion Criteria:

* Disease or serious injury that inhibited participating in the warm-up protocols and subsequent testing sessions.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-10-20 (Actual); Study Completion 2023-10-20 (Actual)

PRIMARY OUTCOMES:
Special judo fitness test (SJFT) | 15 seconds for the 1st set, 30 seconds for sets #2 and #3
  Three sets of time-limited judo throws, assessing the number of throws

SECONDARY OUTCOMES:
Heart rate | During the SJFT, immediately after the SJFT, and 1 minute after the SJFT
  Monitoring of heart rate
Rate of perceived exertion | 30 minutes after each testing session
  Assess perceived exertion

CONTACTS AND LOCATIONS:
Overall Officials: José Afonso, Ph.D., Study Chair — Faculty of Sport of the University of Porto
Locations (1):
- Faculty of Sport of the University of Porto, Porto, Portugal

IPD SHARING:
Plan to Share IPD: Yes
Anonymised data pertaining sample characteristics and results of the implemented assessments will be shared upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Anonymised data pertaining sample characteristics and results of the implemented assessments will be shared upon request. No predicted end date.
Access Criteria: Anonymised data pertaining sample characteristics and results of the implemented assessments will be shared upon request.